CLINICAL TRIAL: NCT00917735
Title: Phase II, Randomized,Double-blind, Placebo-controlled, Study of the Efficacy of Green Tea Extract on Biomarkers of Breast Cancer Risk in High Risk Women With Differing Catechol-O-methyl Transferase (COMT) Genotypes
Brief Title: Green Tea and Reduction of Breast Cancer Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0806M36121; R01CA127236 (NIH)
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Green tea; Breast cancer; Prevention; COMT genotype; EGCG (Epigallocatechin gallate); Mammographic density; Reproductive hormones; IGF axis proteins; Oxidative stress
MeSH Terms: conditions — Breast Neoplasms | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Green tea extract (Experimental): Green tea extract capsules containing 80.7 % total catechins (51.7 % EGCG)
  Interventions: Drug: Green tea extract supplement
- Sugar pill (Placebo Comparator): Placebo capsules containing 50% maltodextrin, 49.5 % cellulose, and 0.5 % magnesium stearate
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Green tea extract supplement — Two green tea extract capsules twice daily after breakfast and dinner for one year
  Other Names: Green tea extract: Corban green tea blend (GTB-3D)
  Arms: Green tea extract
Other: Placebo — Two placebo capsules twice daily after breakfast and dinner for one year
  Other Names: Sugar Pill
  Arms: Sugar pill

SUMMARY:
RATIONALE: Green tea extract contains ingredients (catechins) that may lower the risk of breast cancer.

PURPOSE: This phase II trial is studying how well green tea extract works in preventing breast cancer compared to a placebo in postmenopausal women with high breast density.

The investigators have hypothesized that green tea consumption reduces breast cancer risk, and this effect is seen primarily in women who have the low-activity COMT genotype. The investigators will test this by evaluating the effects of green tea extract on breast cancer biomarkers including mammographic density, plasma insulin-like growth factor 1 (IGF-1), IGF binding protein 3 (IGFBP-3), estrone, estradiol, androstenedione, sex hormone binding globulin (SHBG), urinary estrogen metabolites and plasma F2-isoprostanes.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Primary:

   1.1 To determine the effects of green tea extract consumption (containing 800 mg EGCG per day) for 12 months on the following recognized biomarkers of breast cancer risk:
   1. Mammographic density
   2. Circulating concentrations of insulin-like growth factor 1 (IGF-1) and IGF binding protein 3 (IGFBP-3)
   3. Circulating concentrations of reproductive hormones (estrone, estradiol, androstenedione) and sex hormone binding globulin (SHBG)

   1.2 To determine the effects of COMT genotype on the green tea extract effects described above.
2. Secondary:

2.1 To determine the effects of green tea extract consumption (containing 800 mg EGCG per day) for 12 months on the following hypothesized biomarkers of breast cancer risk:

1. Urinary estrogen metabolites (estrone, estradiol, and their 2-hydroxy, 4-hydroxy, 2-methoxy, and 4-methoxy metabolites, estriol, and 16- hydroxyestrone)
2. Circulating concentrations of F-2 isoprostanes, a recognized biomarker of systemic oxidative stress

2.2 To determine the effects of COMT genotype on the green tea extract effects described above.

2.3 To determine the effects of COMT genotype on catechin metabolism and excretion, as measured by circulating and urinary concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy postmenopausal women aged 50-70 years
* "Heterogeneously dense" (51-75% glandular) or "extremely dense" (>75%glandular) breasts
* Willing to avoid consumption of green tea for 1 year

Exclusion Criteria:

* Positive serological markers of hepatitis B or hepatitis C infections
* Elevated levels of liver enzymes
* Recent (within 6 mo) or current hormone or hormone modification therapy, including systemic hormone replacement therapy, SERMS and aromatase inhibitors
* Current smoker of cigarettes or other tobacco products
* BMI <19 or >40 kg/m2
* Weight change > 10 lbs during the previous year
* History of breast cancer or proliferative breast disease
* Regular consumption of > 7 alcoholic drinks/wk
* Regular consumption of green tea (>1 cup/wk)
* Recent (within 6 mo) or current use of chemopreventive agents such as tamoxifen, raloxifene or aromatase inhibitors
* Participation in any weight loss or weight gain studies
* Currently taking Methotrexate or Enbrel
* History of ovarian cancer
* Any form of cancer in the last 5 years
* Presence of implants

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mindy S Kurzer, Ph.D, Principal Investigator — University of Minnesota
Locations (5):
- United States (5):
  - Fairview Southdale Breast Center, Edina, Minnesota
  - Fairview Maple Grove Breast Center, Maple Grove, Minnesota
  - University of Minnesota Medical Center (UMMC) Breast Clinic, Minneapolis, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Food Science and Nutrition, University of Minnesota, Saint Paul, Minnesota

REFERENCES:
- [Derived] Bathgate JR, Radler DR, Kurzer M, Samavat H. Green tea extract supplementation does not modify plasma concentration of F2-isoprostanes in women who are postmenopause: Findings from a randomized controlled trial. Nutr Res. 2023 May;113:29-38. doi: 10.1016/j.nutres.2023.03.001. Epub 2023 Mar 9. PMID 37011435
- [Derived] Samavat H, Wu AH, Ursin G, Torkelson CJ, Wang R, Yu MC, Yee D, Kurzer MS, Yuan JM. Green Tea Catechin Extract Supplementation Does Not Influence Circulating Sex Hormones and Insulin-Like Growth Factor Axis Proteins in a Randomized Controlled Trial of Postmenopausal Women at High Risk of Breast Cancer. J Nutr. 2019 Apr 1;149(4):619-627. doi: 10.1093/jn/nxy316. PMID 30926986
- [Derived] Arikawa AY, Samavat H, Gross M, Kurzer MS. Plasma F2-isoprostanes Are Positively Associated with Glycemic Load, but Inversely Associated with Dietary Polyunsaturated Fatty Acids and Insoluble Fiber in Postmenopausal Women. J Nutr. 2017 Sep;147(9):1693-1699. doi: 10.3945/jn.117.254631. Epub 2017 Jul 26. PMID 28747487
- [Derived] Samavat H, Newman AR, Wang R, Yuan JM, Wu AH, Kurzer MS. Effects of green tea catechin extract on serum lipids in postmenopausal women: a randomized, placebo-controlled clinical trial. Am J Clin Nutr. 2016 Dec;104(6):1671-1682. doi: 10.3945/ajcn.116.137075. Epub 2016 Nov 2. PMID 27806972
- [Derived] Dostal AM, Arikawa A, Espejo L, Kurzer MS. Long-Term Supplementation of Green Tea Extract Does Not Modify Adiposity or Bone Mineral Density in a Randomized Trial of Overweight and Obese Postmenopausal Women. J Nutr. 2016 Feb;146(2):256-64. doi: 10.3945/jn.115.219238. Epub 2015 Dec 23. PMID 26701796
- [Derived] Dostal AM, Samavat H, Espejo L, Arikawa AY, Stendell-Hollis NR, Kurzer MS. Green Tea Extract and Catechol-O-Methyltransferase Genotype Modify Fasting Serum Insulin and Plasma Adiponectin Concentrations in a Randomized Controlled Trial of Overweight and Obese Postmenopausal Women. J Nutr. 2016 Jan;146(1):38-45. doi: 10.3945/jn.115.222414. Epub 2015 Nov 18. PMID 26581683
- See also: The Minnesota Green Tea Trial (MGTT), a randomized controlled trial of the efficacy of green tea extract on biomarkers of breast cancer risk: study rationale, design, methods, and participant characteristics — http://www.ncbi.nlm.nih.gov/pubmed/26206423
- See also: The safety of green tea extract supplementation in postmenopausal women at risk for breast cancer: results of the Minnesota Green Tea Trial — http://www.ncbi.nlm.nih.gov/pubmed/26051348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2009 through April 2013
Pre-assignment Details: Prior to randomization, participants went through a screening clinic visit in which anthropometric characteristics and blood pressure were measured. In addition, blood was drawn to assess catechol-O-methyltransferase (COMT) genotype, hepatic function, and serological markers of hepatitis B and C virus.
Groups:
- Green Tea Extract: Green tea extract (GTE) supplement: Two green tea extract capsules twice daily after breakfast and dinner for one year. GTE was a decaffeinated green tea extract, and each capsule contained a total of 328.8 ± 28.9 mg catechins including 210.7 ± 11.0 mg of epigallocatechin gallate (EGCG).
- Sugar Pill: Placebo: Two placebo capsules twice daily after breakfast and dinner for one year. Placebo capsules contained maltodextrin, cellulose, and magnesium stearate.
Period: Overall Study
Arm/Group | Green Tea Extract | Sugar Pill
Started | 538 | 537
Completed | 463 | 474
Not Completed | 75 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Green Tea Extract | Sugar Pill | Total
Number analyzed (Participants) | 538 | 537 | 1075
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (5.0) | 59.6 (5.1) | 59.8 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 538 | 537 | 1075
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 516 | 510 | 1026
  Unknown or Not Reported | 17 | 21 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 515 | 505 | 1020
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 538 | 537 | 1075
Height [Mean (Standard Deviation); unit: cm] | 163.5 (6.3) | 164.3 (6.2) | 163.9 (6.2)
Weight [Mean (Standard Deviation); unit: kg] | 67.4 (10.6) | 67.9 (10.5) | 67.4 (10.5)
Waist-to-hip ratio [Mean (Standard Deviation); unit: Ratio] | 0.84 (0.1) | 0.83 (0.1) | 0.83 (0.07)

OUTCOME MEASURES:

1. Primary Outcome: Mammographic Density
Description: Percent mammographic density was measured on digital images using a computer-assisted and quantitative method.
Time Frame: Baseline and month 12
Population: Mammographic density at baseline and month 12
Measure: Geometric Mean (95% Confidence Interval); unit: Percent
Groups:
- Green Tea Extract: Green tea extract (GTE) supplement: Two green tea extract capsules twice daily after breakfast and dinner for one year. GTE was a decaffeinated green tea extract, and each capsule contained a total of 328.8 ± 28.9 mg catechins including 210.7 ± 11.0 mg of EGCG.
Arm/Group | Green Tea Extract | Sugar Pill
Number analyzed (Participants) | 462 | 470
Percent
  Percent mammographic density at baseline | 22.71 [21.39 to 24.10] | 21.84 [20.59 to 23.17]
  Percent mammographic density at month 12 | 22.09 [20.77 to 23.50] | 21.13 [19.88 to 22.47]

2. Primary Outcome: Circulating Concentrations of Reproductive Hormones Including Estrone, Estradiol, Androstenedione, Testosterone, and Sex Hormone Binding Globulin (SHBG)
Description: Circulating levels of reproductive hormones including estrone, estradiol, androstenedione, testosterone and SHBG were measured in fasting blood samples by liquid chromatography/tandem mass spectrometry method.
Time Frame: Baseline and month 12
Population: Circulating concentrations of reproductive hormones including estrone, estradiol, androstenedione, testosterone, sex hormone binding globulin (SHBG) at baseline and month 12
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Green Tea Extract | Sugar Pill
Number analyzed (Participants) | 463 | 474
pg/ml
  Circulating estrone at baseline | 22.8 [21.6 to 24.0] | 23.6 [22.4 to 24.9]
  Circulating estrone at month 12 | 22.5 [21.3 to 23.7] | 22.4 [21.3 to 23.6]
  Circulating estradiol at baseline | 3.4 [3.1 to 3.8] | 3.7 [3.3 to 4.1]
  Circulating estradiol at month 12 | 3.7 [3.4 to 4.1] | 3.1 [2.8 to 3.5]
  Circulating androstenedione at baseline | 479.8 [459.4 to 501.2] | 507.2 [485.9 to 529.5]
  Circulating androstenedione at month 12 | 468.8 [450.2 to 488.3] | 479.5 [460.6 to 499.1]
  Circulating testosterone at baseline | 151.0 [142.7 to 159.7] | 161.6 [152.8 to 170.8]
  Circulating testosterone at month 12 | 158.1 [149.9 to 166.9] | 155.1 [147.1 to 163.6]
  Circulating SHBG at baseline | 68.1 [65.0 to 71.3] | 69.1 [66.0 to 72.3]
  Circulating SHBG at month 12 | 68.7 [65.5 to 72.0] | 68.7 [65.5 to 72.0]

3. Primary Outcome: Circulating Concentrations of IGF Axis Proteins Including IGF-1 and IGFBP-3
Description: Circulating levels of IGF-1 and IGFBP-3 were measured in fasting blood samples by ELISA method.
Time Frame: Baseline and month 12
Population: Circulating concentrations of IGF axis proteins including insulin-like growth factor (IGF-1) and IGF binding protein 3 (IGFBP-3) at baseline and month 12
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Green Tea Extract | Sugar Pill
Number analyzed (Participants) | 462 | 473
ng/ml
  Circulating IGF-1 at baseline | 87.5 [85.3 to 89.8] | 88.3 [86.1 to 90.5]
  Circulating IGF-1 at month 12 | 83.7 [81.6 to 85.8] | 83.1 [81.0 to 85.2]
  Circulating IGFBP-3 at baseline | 2048.0 [2008.9 to 2088.0] | 2047.6 [2008.9 to 2087.1]
  Circulating IGFBP-3 at month 12 | 2048.1 [2008.0 to 2089.1] | 2040.7 [2001.0 to 2081.0]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse event information was coded and graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.
Arm/Group | Green Tea Extract | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 12/538 | 8/537
Other Adverse Events (participants affected / at risk) | 407/538 | 391/537
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Green Tea Extract (N=538) | Sugar Pill (N=537)
Elevated ALT or AST enzyme (Hepatobiliary disorders) | 7 (9) | 0 (0)
Motorcycle accident (Social circumstances) | 0 (0) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Social circumstances) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 3 (3) | 2 (2)
Acoustic Neuroma (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diagnosis of Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Green Tea Extract (N=538) | Sugar Pill (N=537)
Nausea (Gastrointestinal disorders) | 235 (235) | 184 (184)
Infections (Infections and infestations) | 216 (216) | 217 (217)
Vascular (Vascular disorders) | 154 (154) | 144 (144)
Respitory (Respiratory, thoracic and mediastinal disorders) | 122 (122) | 122 (122)
General (General disorders) | 69 (69) | 77 (77)
Musuclar (Musculoskeletal and connective tissue disorders) | 65 (65) | 69 (69)
Other (General disorders) | 280 (280) | 218 (218)

LIMITATIONS AND CAVEATS:
We had limited success in recruiting minority populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No